CLINICAL TRIAL: NCT00600691
Title: The Use of Finasteride to Reduce Hematuria and Hematospermia Following TRUS Prostate Biopsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not achieve enrollment goal and decided to terminate early
Sponsor: University of British Columbia (Other)
Collaborators: Health Canada (Other Government); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H07-01188; Health Canada Control #118638; Merck Frosst #IISP #P2587
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Hematuria; Hematospermia
Keywords: Finasteride; hematuria; hematospermia; prostate biopsy
MeSH Terms: conditions — Hematuria; Hemospermia | interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 5mg finasteride orally, daily for 2 weeks prior to prostate biopsy and one week following prostate biopsy.
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride — one tablet (5mg) of finasteride

SUMMARY:
The purpose of our study is primarily to evaluate the effects of 5mg finasteride on hematuria and hematospermia commonly associated with prostate biopsies. We hypothesize that 5mg of finasteride daily for two weeks preceding TRUS prostate biopsy and one week following will reduce hematuria and hematospermia commonly seen as complications following prostate biopsy. We also hypothesize that reducing complications will decrease concern among subjects and make for a more tolerable overall procedure than compared with subjects treated with placebo.

DETAILED DESCRIPTION:
Study Purpose:

The purpose of our study is primarily to evaluate the effects of 5mg finasteride on hematuria and hematospermia commonly associated with prostate biopsies. We will also examine how effective the dosing of finasteride administered two weeks prior to biopsy and one week following. We will also use the subject questionnaire to assess subject's attitudes and concerns about hematuria and hematospermia. We will examine the overall subjective tolerability of the biopsy procedure, concerns about sexual function, anxiety surrounding prostate cancer, and urination following the procedure. Questionnaires will use a 10 point visual analog scale to gauge subject's attitudes and concerns. We will examine for any statistically significant correlations between these parameters and the complications we are monitoring. We will also monitor side effects of subjects, in an effort to gauge the potential risks associated with short term usage of finasteride compared to any benefits afforded by finasteride on reducing hematuria and hematospermia.

Hypotheses:

Based on the previous research into the molecular mechanisms of finasteride, we hypothesize that 5mg of finasteride daily for two weeks preceding TRUS prostate biopsy and one week following will reduce hematuria and hematospermia commonly seen as complications following prostate biopsy. We also hypothesize that reducing complications will decrease concern among subjects and make for a more tolerable overall procedure than compared with subjects treated with placebo.

Objectives:

To determine the effectiveness of 5mg finasteride administered two weeks prior to prostate biopsy and one week following on reducing hematuria and hematospermia following biopsy.

To gauge subject's concerns relating to hematuria, hematospermia, and transmitting prostate cancer to partners following TRUS prostate biopsy.

To examine subject's subjective sexual function and urination in relation to their treatment group.

To demonstrate benefits of finasteride in relation to the safety and tolerability of treatment.

Endpoints:

Differences in rate and severity of hematuria and hematospermia among subjects in treatment and placebo groups.

Differences in complications following biopsies, such as hospitalization and requirement for blood transfusion, between treatment and placebo groups.

Differences between placebo group and finasteride treatment group in: overall subjective experience of biopsy procedure, concern relating to hematuria and hematospermia, sexual function, and urination following prostate biopsy.

Monitor side effects between placebo and finasteride when administered for three weeks total duration.

Research design:

The study we plan to conduct will be a randomized, double-blind, placebo controlled study to determine the effects of 5mg finasteride on the rate/severity of hematuria and hematospermia following TRUS prostate biopsy.

A total of 50 subjects will be randomized into one of two groups. One group will receive 5mg of finasteride orally for two weeks prior to TRUS biopsy, and one week after the biopsy. Another group will receive a placebo orally for two weeks prior to the procedure and one week following the biopsy. Patients will be identified for participation by existing indication for TRUS prostate biopsy, and subsequently enrolled. Subjects will receive the current standard of care in addition to participating in this study.

The study is designed to investigate the effects of finasteride compared to placebo on hematuria and hematospermia following prostate biopsy. Subjects will be assigned to treatment groups using a randomization process to eliminate selection bias, and to ensure that any differences between the two study groups are due to random chance. The study has been designed as placebo controlled and double blinded to ensure that investigator and subject ascertainment biases are minimized. As there is no current prophylactic or other treatment to decrease the rate/severity of hematuria and hematospermia following prostate biopsies, this does not raise any ethical concerns in the placebo group.

Subject recruitment will be done on an ongoing basis.

Statistical analysis plan:

We will perform statistical analysis on the data collected from this study. We will examine whether there is a statistically significant difference in the rates of hematuria and hematospermia between placebo and finasteride treatment groups. We will also examine for any statistically significant relationships between study groups (placebo versus finasteride) and concern regarding hematuria/hematospermia, satisfaction with/tolerability of the biopsy, concern with prostate cancer transmission, sexual/urinary function, and side effects.

Research Procedures:

Subjects will be identified as potential participants for this study in the office of Dr. Pommerville. Dr. Pommerville will identify subjects from within his urology practice as needing a TRUS biopsy out of medical necessity for reasons unrelated to enrollment in this study. The indications for prostate biopsy are usually based on clinical suspicion using a combination of digital rectal examination and prostate specific antigen blood testing. Once identified as potential candidates for participation in this study, Dr. Pommerville will give the potential subject a detailed explanation of the study and will explain the content in the informed consent form. Once the patient has read the consent form and understands what the study entails, they will make a decision whether or not to enroll in this study. Once informed consent has been obtained, subjects will be assigned a unique identification number, which will not be used for any other purposes. This identification code will have features that allow the code to be broken in an emergency situation. At this time, subjects will be randomly assigned to the placebo or treatments groups in a double blind fashion.

Subjects will be given a three week supply of 5mg of finasteride or placebo and detailed instructions on how they are to take their medication/placebo. They will be instructed to take their medication/placebo, one tablet (5mg) of finasteride/placebo orally each day for two weeks prior to biopsy and one week following. This will be in addition to the standard of care that is normally given with prostate biopsy (antibiotics, enema). They will be given an appointment to undergo prostate biopsy in two weeks. Subjects will be instructed that if they decide to withdraw from this study, they may do so at any time, and return the unused medication to Dr. Pommerville's office at follow up

Subjects will then undergo TRUS prostate biopsy two weeks later as part of their standard medical care at either the Royal Jubilee Hospital or Victoria General Hospital. Equipment and procedures will not differ between these sites. Patients will be followed up at this point by Dr. Pommerville on their participation and adherence to study protocol. If subjects have not been compliant with the protocol, they will be withdrawn from the study. Subjects will receive repeat instructions on taking their medication and released as would be expected as part of the standard of care for prostate biopsies. They will be given an appointment for two weeks from the TRUS biopsy to see Dr. Pommerville in his clinic. They will be reminded to come to the clinic approximately 20 minutes prior to their appointment time so that Nathan Hoag (Medical student) may administer a questionnaire in accordance with what was described to them by the informed consent form.

Subjects will present for their scheduled two week follow up appointment to Dr. Pommerville's office. This practice is in accordance with the normal standard of care. Nathan Hoag will administer the subject questionnaire at this point. Questionnaires will be administered prior to subjects seeing Dr. Pommerville for biopsy results in an effort to minimize emotional influence on the results of the questionnaire. This is the last visit in the standard medical care for prostate biopsy. Subjects are instructed to follow up with Dr. Pommerville or their family physicians should they have additional concerns. At this time, subjects will be reminded that they are to return to Dr. Pommerville's office in an additional two weeks, where the medical student will administer the questionnaire for a second time to monitor any ongoing changes (4 weeks since procedure).

In addition to the patient questionnaire, previously described grading systems will be used to quantify the incidence and severity of hematuria and hematospermia among subjects at two and four weeks.18,19 Hematospermia grading systems quantify hematospermia as mild (less than 7 days), moderate (7 to 14 days), and severe (more than 14 days). Hematuria is defined as grossly passing blood or blood clots in the urine. Hematuria is stratified using minor episodes (lasting 24 hours or less), moderate episodes (lasting more than 24 hours, but not requiring hospital admission), and severe episodes (clot retention and hospital admission). Hematuria will then be graded according to the following system: grade 0 (no gross hematuria), grade 1 (up to 2 minor episodes or 1 moderate episode), grade 2 (more than 2 minor episodes or 1 moderate episode), grade 3 (1 or more severe episodes).

This will be the conclusion of the study for subjects. They will be reminded that they are free to contact Nathan Hoag should they have any concerns or questions. They will also be reminded that they may follow up with Dr. Pommerville or their family physicians should they need to.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to the participation in any study related activity.
2. Male subject already identified as requiring TRUS prostate biopsy for unrelated medical reasons.

Exclusion Criteria:

1. Suspected or known liver disease.
2. Suspected or known hematological disorders.
3. Subjects who are candidates for immediate surgery.
4. Known hypersensitivity to any component of the product.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Differences in rate and severity of hematuria and hematospermia among subjects in treatment and placebo groups. | 2 & 4 weeks

SECONDARY OUTCOMES:
Differences between placebo group and finasteride treatment group in: complication rates, overall subjective experience of biopsy procedure, and concern relating to biopsy. Monitor side effects between placebo and finasteride. | 2 & 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pommerville, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia